CLINICAL TRIAL: NCT04381182
Title: Impact of Heart Rate Variability Modulation on Stress and Performance Among Neurosurgical Residents
Brief Title: Heart Rate Variability and Stress Management Enhancement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient data/adherence
Sponsor: Joseph Maroon (Other)
Collaborators: Apollo Neuro (Unknown)
Responsible Party: Sponsor-Investigator, Joseph Maroon, Clinical Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY19020291
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Stress; Heart Rate Variability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biostrap/Apollo Device Use (Other): Participants wear a Biostrap wearable device which measures steps, heart rate, heart rate variability, sleep metrics, and quantitative data in typical day-to-day activities of residents. Participants then again wear Biostrap except now also with the Apollo device which is worn around the ankle and is suggested to modulate heart rate variability and perceived stress of participants.
  Interventions: Device: Apollo Wearable Device

INTERVENTIONS:
Device: Apollo Wearable Device — Participants wear Apollo device which generates vibration frequencies on skin and can be controlled by the user

SUMMARY:
This study will be conducted by using two devices (Apollo and Biostrap) for monitoring of baseline physiologic variables and heart rate variability. The biostrap will be worn by residents and will monitor heart rate, heart rate variability, respiratory rate, sleep patterns, steps, etc. The Apollo is a pulse generator device aimed at modulating heart rate variability for (hopefully) reduction in stress and improving performance in and around the hospital. Resident neurosurgeons will wear the biostrap for a two week cycle and follow that with the addition of the Apollo device for heart rate variability modulation.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical Resident (UPMC)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline to two month heart rate variability | Baseline, Two Month. Analyzed via paired t-test and assessing change between each outcome time point
  Quantitative (average range, beats per minute)
Change from baseline to two month Perceived Stress Scale | Baseline, Two Month. Analyzed via paired t-test and assessing change between each outcome time point
  Questionnaire, 14 point form/scale ranging from 0-50 with higher scores signifiying increased stress
Change from baseline to two month Quick Inventory of Depressive Symptomatology (QIDS) | Baseline, Two Month. Analyzed via paired t-test and assessing change between each outcome time point
  Questionnaire ranging from 0-27 and measuring major depressive symptomatology. Higher scores signify more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Maroon, Principal Investigator — Department of Neurological Surgery
Locations (1):
- UPMC Presbyterian Hospital Department of Neurological Surgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified changes in heart rate variability, de-identified changes between QIDS and PSS questionnaires.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available at one month from study start and will be available for two months from study start.
Access Criteria: Principal investigator and three additional primary study members will have access to data.